CLINICAL TRIAL: NCT02640508
Title: Phase II Trial of Eribulin and Lenvatinib in Advanced Solid Tumors (CTMS# 15-2139)
Brief Title: Eribulin and Lenvatinib in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia G. Kaklamani (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Virginia G. Kaklamani, Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 15-2139; HSC20150891H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2015-11-26; First posted 2015-12-29 (Estimated); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — eribulin; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Eribulin and lenvatinib (Experimental): Eribulin will be given on days 1 and 8. Lenvatinib will be given daily in each 28 day cycle.
  Interventions: Drug: Eribulin; Drug: Lenvatinib

INTERVENTIONS:
Drug: Eribulin — Will be given by I.V. at 1.4 mg/m2 on day 1 and day 8.
  Other Names: Halaven
Drug: Lenvatinib — Will be taken orally at 20-24 mg daily in each 21 day cycle.
  Other Names: Lenvima

SUMMARY:
The overall purpose of this study is to determine the overall response rate, efficacy and safety of the combination of eribulin and Lenvatinib.

DETAILED DESCRIPTION:
This is a phase II clinical trial of the combination of eribulin, and Lenvatinib. A cycle will be defined as 21 days. Eribulin will be given on days 1 and 8 of each cycle. Lenvatinib will be given daily during each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV breast cancer, stage IV NSCLC (Non-Small Cell Lung Cancer) (, stage IV sarcoma
* ECOG (Eastern Cooperative Oncology Group) PS (Performance Status) 0-2
* Measurable disease
* No more than 4 prior chemotherapeutic regimens for metastatic disease
* Patients must be >/= 18 years.
* Patients may not have received eribulin or lenvatinib previously
* Patients must have a life expectancy of greater than 12 weeks.
* Patients may have had a prior diagnosis of cancer if it has been > 5 years since their last treatment and are considered free of disease.
* Patients must have normal organ and marrow function as defined below:

Leukocytes ≥ 3,000/uL Absolute neutrophil count ≥ 1,500/uL Platelets ≥ 100,000/uL Child Pugh score ≤ 10 Patients must be able to swallow and retain oral medication. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Women who are pregnant or lactating are not eligible for study treatment.
* Patients who are undergoing concomitant radiotherapy are NOT eligible for participation.
* Patients who are receiving any other investigational agents or concurrent anticancer therapy are NOT eligible for participation. Previous systemic treatment and/or radiation therapy is allowed with a 14 day washout period prior to registration.
* Lesions that have been radiated previously cannot be considered target lesions
* Prior treatment related side effects must have resolved to < Grade 2 severity per Common Terminology Criteria for Adverse Events (CTCAE version 4.03), except alopecia and infertility.
* Patients who are taking any herbal (alternative) medicines are NOT eligible for participation. Patients must be off any such medications by the time of registration.
* Patients with known brain metastases are NOT eligible for participation unless the brain metastases are treated (either with surgical excision, stereotactic radiosurgery or radiotherapy) and have been stable for at least 4 wks per MR performed, the patient is asymptomatic and has discontinued corticosteroids if taken for that purpose.
* Patients with any of the following conditions or complications are NOT eligible for participation:

  1. GI tract disease resulting in an inability to take oral medication
  2. Malabsorption syndrome
  3. Require IV alimentation
  4. History of prior surgical procedures affecting absorption
  5. Uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
  6. Hypersensitivity of any of the components of eribulin or lenvatinib
  7. History of significant neurological ( no neuropathy more than grade 2) or psychiatric disorders
  8. Significant non neoplastic liver disease (Cirrhosis, active chronic hepatitis)
  9. Immunocompromised subjects, including patients with human immunodeficiency virus
  10. Significant non neoplastic renal disease
  11. Active infection requiring systemic therapy.
  12. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment
  13. Prolongation of QTc interval to more than 480 milliseconds when electrolyte balance is normal
  14. Major surgery within 4 weeks prior to first dose of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05; Primary Completion 2020-11-24 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy and Research Center University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with the following diagnoses will be included: metastatic solid tumors including breast cancer, NSCLC and soft-tissue sarcoma.
Pre-assignment Details: A 10-patient safety run-in phase for each drug combination will be conducted during cycle 1 of the treatment and subjects evaluated with the remainder of subjects enrolled. After the first 10 subjects have been enrolled the phase II enrollment will begin with the aim of enrolling an additional 20 subjects. All surviving subjects who received study drug will be followed for disease progression and survival. Evaluation of the subjects will be conducted as a single group.
Groups:
- Lenvatinib and Eribulin: Eribulin will be administered on cycle days 1 and 8; Lenvatinib is an orally administered medication given daily throughout each cycle. On days when both drugs are administered, Eribulin will be administered immediately prior to Lenvatinib.
Period: Overall Study
Arm/Group | Lenvatinib and Eribulin
Started | 29
Escalation to Higher Dose | 0
Completed | 0
Not Completed | 29
Not completed — Death | 19
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Eribulin and Lenvatinib
Number analyzed (Participants) | 29
Age, Continuous [Median (Standard Deviation); unit: years] | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
ECOG performance status [Number; unit: Percentage] — Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 life expectancy of greater than 12 weeks, and adequate hematologic, liver and renal function.
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  Percentage
    0 | 17
    1 | 9
    2 | 3
Tumor history [Count of Participants; unit: Participants]
  Mammary carcinoma | 17
  Lung carcinoma | 6
  Sarcoma | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Lenvatinib and Eribulin (Phase II)
Description: Defined as the percentage of patients with best overall response of complete response (CR) or partial response (PR) as assessed by independent imaging review.
Time Frame: The overall response rate will be assessed after two cycles of therapy (1 cycle = 3 weeks) until the date of first documentation of disease progression or death (whichever occurs first) over an average of 18 months.
Population: Only 23 patients had evaluable disease as 6 subjects came off study early prior to first assessment due to toxicities.
Measure: Number; unit: participants
Arm/Group | Combination Eribulin and Lenvatinib
Number analyzed (Participants) | 23
participants
  Partial Response | 7
  Stable Disease | 13
  Progression of Disease | 3

2. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) will be defined as the time from the first study treatment to the first occurrence of progression or death.
Time Frame: Baseline to 50 months
Measure: Median (Full Range); unit: months
Arm/Group | Combination Eribulin and Lenvatinib
Number analyzed (Participants) | 23
months | 7.4 [1 to 47]

3. Secondary Outcome: Overall Survival Rate
Time Frame: Baseline to 50 months
Measure: Median (Full Range); unit: Months
Arm/Group | Combination Eribulin and Lenvatinib
Number analyzed (Participants) | 23
Months | 8.2 [1 to 47]

4. Secondary Outcome: Lenvatinib and Eribulin Toxicities Will be Graded Using NCI CTCAE Version 4.03
Description: Adverse events are graded in the NCI CTCAE version 4.03 scale and reported by number of adverse events per grade
Time Frame: Safety will be evaluated from the time of registration until 30 days after last dose of treatment, resolution of the related AE or death up to 40 months.
Population: All subjects that received investigational product, including those from Phase 1 that were not included in the analysis of data
Measure: Number; unit: Events
Arm/Group | Combination Eribulin and Lenvatinib
Number analyzed (Participants) | 29
Events
  Grade 1 | 182
  Grade 2 | 130
  Grade 3 | 57
  Grade 4 | 9
  Grade 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all subjects from first cycle of the administration of the study drug through the end of the active study follow-up of the study during treatment up to 50 months. No subjects were escalated to a higher dose due to toxicity concerns, so all participants received the same dose.
Groups:
- Combination Eribulin and Lenvatinib: Eribulin will be given on days 1 and 8. Lenvatinib will be given daily in each 28 day cycle.
  For each cycle: Eribulin: Will be given by I.V. at 1.4 mg/m2 on day 1 and day 8 and Lenvatinib: Will be taken orally at 20-24 mg daily days 1-21 of each 28 day cycle.
Arm/Group | Combination Eribulin and Lenvatinib
All-Cause Mortality (participants affected / at risk) | 19/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Eribulin and Lenvatinib (N=29)
Neutrophil count decreased (Blood and lymphatic system disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Epistaxis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Myalgia (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Palmar-plantar erthrodysestesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Eribulin and Lenvatinib (N=29)
Oral mucositis (Gastrointestinal disorders) | 18 (32)
Fatigue (General disorders) | 16 (23)
Neutrophil count decrease (Blood and lymphatic system disorders) | 10 (25)
Nausea (Gastrointestinal disorders) | 14 (16)
Vomiting (Gastrointestinal disorders) | 10 (13)
Hypertension (Cardiac disorders) | 8 (16)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Gastrointestinal disorders) | 6 (6)
Hypothyroidism (Endocrine disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Decreased platelet count (Blood and lymphatic system disorders) | 4 (4)
Decreased white blood cell count (Blood and lymphatic system disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine Amino transferase increased (Hepatobiliary disorders) | 3 (3)
Alkaline Phosphatase increased (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 3 (4)
Increased bilirubin (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1) — Taste disorder
Dyspepsia (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02640508/Prot_SAP_000.pdf